CLINICAL TRIAL: NCT05707494
Title: A Multicenter Prospective Observational Study With a Control Group to Evaluate the Efficacy and Safety of LPS Adsorption Using the Efferon LPS NEO Device in Children With SepSis (LASSO NEO).
Brief Title: Lipopolysaccharide Adsorption (Efferon LPS NEO) in Children With Sepsis
Acronym: LASSONEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Collaborators: Ligand Research, LLC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-lps-2023-01
Record Dates: First submitted 2023-01-20; First posted 2023-02-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Septic Shock
Keywords: septic shock; sepsis; extracorporeal therapy; LPS adsorption
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: A multicenter prospective observational study with a control group to evaluate the efficacy and safety of LPS Adsorption using the Efferon LPS NEO device in children with SepSis (LASSO NEO).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic therapy + Efferon LPS NEO (Experimental): Study group: Basic therapy + Efferon LPS NEO - 32 patients, prospective enrollment.
  Interventions: Device: Efferon LPS NEO
- Baseline therapy (No Intervention): Control group: Basic therapy - 46 patients, retrospective enrollment. Basic therapy is the routine practice of the institution for the treatment of patients with sepsis (conservative anti-infective therapy). Antibacterial therapy regimens, antibiotic dosage adjustment regimens for AKI and prolonged RRT procedures are not specifically prescribed in the CT Plan.

INTERVENTIONS:
Device: Efferon LPS NEO — Efferon LPS NEO, a medical device, which is a cylindrical body filled with a polymeric hemosorbent that selectively absorbs LPS and excess cytokines. The device is used for extracorporeal therapy to relieve septic shock in the treatment of sepsis.
  Arms: Basic therapy + Efferon LPS NEO

SUMMARY:
One of the major health problems in the world is sepsis, the number of cases of which, according to WHO, annually reaches 20-30 million. The decrease in the sensitivity of bacterial pathogens to antibiotics, the widespread use of invasive diagnostic and treatment methods, the increased role of opportunistic microorganisms and fungi, and the increase in the number of people with severe chronic diseases led to an increase in the incidence of sepsis in the period from 1979 to 1979. 2000 by 8.7% per annum.

Sepsis is one of the leading causes of hospital mortality in children. Multicenter cross-country studies of pediatric sepsis using a prospective methodology in nearly 7,000 children (mean age 3 years) in 128 pediatric intensive care units (ICUs) in 26 different countries showed that a typical 16-bed intensive care unit should have, on average, at least one child with sepsis.

Sepsis and septic shock in most cases are accompanied by the development of multiple organ failure syndrome (MODS). The frequency of adverse outcomes directly depends on the number of organ systems involved in MODS: it increases from 6% in patients with dysfunction of one organ at the time of admission to the intensive care unit to 65% in patients with organ failure of 4 systems or more. Despite modern advances in resuscitation and antimicrobial chemotherapy, if the etiological agent of sepsis is gram-negative flora, mortality can reach 75%.

Numerous studies have shown that the use of extracorporeal sorption methods that eliminate endotoxin improves the results of treatment of patients with septic shock. The use of LPS selective adsorption is both an etiological and pathogenetic method of treatment, which justifies the need for its use in the complex intensive care of sepsis and septic shock.

The method of hemosorption technology using a cartridge based on a mesoporous supercrosslinked copolymer of styrenedivinylbenzene with an LPS-selective ligand immobilized on the surface, which has the ability to neutralize the biological activity of endotoxin by binding lipid A, the main pathogenic site of LPS. the molecule matters.

The main goal of the study was to obtain data on the efficacy and safety of using the Efferon LPS NEO hemosorption column for the adsorption of lipopolysaccharides during extracorporeal detoxification in children aged 1 month to 14 years with sepsis.

DETAILED DESCRIPTION:
One of the major health problems in the world is sepsis, the number of cases of which, according to WHO, annually reaches 20-30 million. Decreased sensitivity of bacterial pathogens to antibiotics, widespread use of invasive methods of diagnosis and treatment, increased role of opportunistic microorganisms and fungi, increased the number of people with severe chronic diseases led to an increase in the incidence of sepsis in the period from 1979 to 2000 by 8.7% annually.

Sepsis is one of the leading causes of hospital mortality in children. Multicenter studies in pediatric sepsis in various countries using a prospective methodology in nearly 7,000 children (mean age 3 years) in 128 pediatric intensive care units (ICUs) in 26 different countries showed that in a typical 16-bed PICU, on average there must be at least one child with sepsis.

In the United States, 75 thousand cases of sepsis in children are recorded annually, and the mortality rate for severe sepsis is 21%. Importantly, nearly 25% of sepsis survivors had a clinically significant health-related deterioration in quality of life, with one in three survivors being discharged with a disability (24% of previously healthy children were discharged with some form of disability).

In a recent systematic review and meta-analysis of the epidemiology of sepsis, the incidence of sepsis in children was 48 cases per 100,000 people per year, and septic shock was 22 cases per 100,000 people per year. In general, the authors determined the incidence of 1.2 million cases of sepsis in children per year. Mortality in children with septic shock ranged from 9 to 20%. Significantly, this systematic review did not include studies from low-income countries where morbidity and mortality from sepsis in children is likely to be higher.

Sepsis and septic shock in most cases are accompanied by the development of multiple organ failure syndrome (MODS). The frequency of adverse outcomes directly depends on the number of organ systems involved in MODS: increasing from 6% in patients with dysfunction of one organ at the time of admission to the ICU to 65% in patients with organ failure of 4 systems or more. Also, lethality is largely determined by the etiology of this complication. Despite modern advances in antimicrobial chemotherapy, if the etiological agent of sepsis is gram-negative flora, mortality can reach 75% and the overall prognosis of patients with endotoxemia and septic shock remains extremely poor.

Hemosorption is a method of extracorporeal removal of toxic substances from the blood by their sorption on a porous material. Hemosorption can be a good addition or replacement for classical methods of hemofiltration and hemodialysis, if the diffusion or convection of toxic substances through the membrane is not efficient enough.

Currently, with the help of hemosorbents based on highly cross-linked styrene/divinylbenzene copolymers, it is possible to remove endo- and exotoxins of acute and chronic renal and hepatic failure, eliminate intoxication with pharmacological drugs, drugs and poisons, and also remove cytokines that are formed in excess during sepsis and systemic inflammatory syndromes. other etiology.

Numerous studies have shown that the use of extracorporeal sorption methods that eliminate endotoxin improves the results of treatment of patients with septic shock. The use of selective LPS adsorption is both an etiological and pathogenetic method of treatment, which justifies the need for its use in the complex intensive care of sepsis and septic shock.

Hemosorption is indicated in patients who suffer from sepsis and are in a state of sepsis-induced hypotension or "warm shock" despite adequate treatment of the primary site of infection. The use of hemosorption should be considered justified if there is a threat of developing sepsis and septic shock, even in the absence of obvious signs of MODS. At the same time, it is difficult to have an accurate idea of the level of endotoxin in the patient's blood before conducting selective liposaccharide sorption due to the methodological difficulties of accurately express determination of the level of LPS in the blood.

Timely application of the method of multimodal (lipopolysaccharide and cytokine) HP will reduce the mortality of patients and the number of antibacterial drugs and drugs used to treat MODS, as well as the length of stay in the ICU and the duration of hospitalization in general.

The main purpose of this non-interventional study is to obtain data on the efficacy and safety of using the Efferon LPS NEO medical device for lipopolysaccharide adsorption during extracorporeal detoxification in children aged 1 month to 14 years with sepsis.

The method of hemosorption technology using a cartridge based on a mesoporous supercrosslinked styrene-divinylbenzene copolymer with an LPS-selective ligand immobilized on the surface, which has the ability to neutralize the biological activity of endotoxin by binding lipid A, the main pathogenic site of the LPS molecule, has been especially relevant in the last 10 years.

Endotoxin, one of the most potent mediators of sepsis, is found in high concentrations in approximately 50% of patients with septic shock. Numerous trials have shown that the use of endotoxin-eliminating extracorporeal sorption techniques improves outcomes in patients with septic shock.

In patients treated with hemosorption therapy, a rapid improvement in the state according to the SOFA scale was noted, which led to a decrease in the length of stay in the ICU compared with patients in the control group. A systematic clinical review of 978 cases showed that mortality among patients treated with GP using a polymyxin cartridge in addition to conventional treatment was 33.5% compared with 61.5% in the control group receiving only conservative anti-infective therapy.

The EUPHAS study, which included 64 patients, showed that the use of the method of selective sorption of endotoxin using a polymyxin B cartridge can increase 28-day survival from 47 to 68%, and in-hospital survival from 33 to 59%, i.e., it makes it possible to reduce mortality in patients with sepsis and septic shock almost 2 times.

Despite the widespread use in recent years of methods for hemosorption of LPS and cytokines, there are no developed protocols for this type of therapy for pediatric patients.

Efferon LPS NEO (Efferon Company, Moscow, Russia) is a device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by selective adsorption of lipopolysaccharides (bacterial endotoxins) and non-selective adsorption of cytotoxins with a molecular size of up to 55 kDa (multimodal sorption).

Differences of the multimodal GP method:

1. the ability to effectively deal with endotoxemia and nonspecific inflammatory process;
2. the ability to prevent severe complications and organ damage and increase survival;
3. the ability to control the course of treatment and quickly respond to changes in the patient's condition (in contrast to the use of traditional antibacterial drugs);
4. the ability to significantly reduce the cost of pharmacotherapy and other methods of treatment, avoid wasteful costs and reduce the length of stay of patients in the ICU with an overall increase in survival compared to traditional antimicrobial therapy.

Efferon LPS NEO is a cylindrical polycarbonate body filled with spherical granules of LPS-selective hemosorbent and isotonic sodium chloride solution. The device is manufactured according to TU 32.50.50-001-12264678-2018, has passed the necessary tests and is registered in Russia as a medical device RZN 2019/8886 of 06/27/2022.

ELIGIBILITY:
Inclusion Criteria:

* Weight from 5 kg. up to 40 kg (main criterion),
* Age from 1 month to 14 years,
* No more than 12 hours from the moment of establishment of DZ - Sepsis in accordance with the criteria of SEPSIS-3 (2016, modified for childhood), most likely, Gr-etiology, at the time of inclusion.
* The immediate postoperative period in case of abdominal nature of sepsis (no more than 12 hours after surgery),
* If the patient has a focus of surgical infection, then it should be sanitized,
* pSOFA scale ≥ 6 points, or an increase in negative dynamics on the pSOFA scale by 2 or more points over 12 hours of observation,
* The patient's condition allows for therapy with the Efferon LPS NEO column for at least 4 hours.

Exclusion Criteria:

* Weight below 5 kg and over 40 kg,
* Age less than 1 month and over 14 years old,
* Failure to obtain informed consent from the patient's parents, family member or legal representative,
* The presence of a focus of non-sanitized surgical infection,
* Use in the treatment of other methods of extracorporeal removal of LPS and inflammatory mediators (hemofilters with highly permeable and surface-modified membranes),
* Acute pulmonary embolism,
* Intracranial hemorrhage or bleeding tendency in general,
* Induced aplasia of hematopoiesis,
* If it is impossible to provide vascular access necessary for the method,
* Any other condition that, in the opinion of the Investigator, would prevent the patient from being a suitable candidate for inclusion in the trial (for example, a chronic disease in the terminal stage or a mental disorder that affects the methodology for conducting a hemoperfusion procedure, as well as for patients who have a "palliative status ").

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of Efferon LPS NEO Hemoperfusion on pSOFA (pediatric Sequential Organ Failure Assessment) Scores in Patients with Sepsis | 1-7 days
  The value of indicators on the pSOFA scale every 24 hours ± 1 hour from the start of hemoperfusion (0 hour) to 7 days. The pSOFA score was developed using validated age-adjusted cut points for the cardiovascular and renal criteria from the second Pediatric Logistic Organ Dysfunction (PELOD-2) scoring system. Scores were calculated daily from admission to the PICU until day 7 of stay, discharge, or death, whichever came first.The pSOFA index is equal to the sum of six indicators. The higher the score, the greater the insufficiency of the system being assessed. The higher the overall index, the greater the degree of multiorgan dysfunction. Violation of the function of each organ (system) is assessed separately in dynamics against the background of intensive therapy. The lower the pSOFA index, the less pronounced organ failure and the better the patient's survival prognosis.

SECONDARY OUTCOMES:
Effect of Efferon LPS NEO hemoperfusion on systemic hemodynamic parameters after initiation of use in patients with sepsis complicated by septic shock | 1-72 hours
  Duration (hours) of vasopressor and inotropic support (where applicable)
Influence of hemoperfusion Efferon LPS NEO in extracorporeal therapy of patients with complicated sepsis septic shock | 1-14 days
  Time (number of days) from enrollment in the study to the earliest point at which "resolution of septic shock" is achieved. Event criteria: 1) cessation of vasopressor support (maintained effect for 4 hours) and 2) Investigator scores as "resolved" from baseline to day 14 or hospital discharge (if discharge occurs before day 14)
Effect of LPS NEO Efferon hemoperfusion on endotoxin activity | 1-72 hours
  Value of endotoxin levels every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours
Effect of the Efferon LPS NEO hemoperfusion on pulmonary oxygen metabolism function | 1-72 hours
  Value of oxygenation index (Pa02 / Fi02 (Pa) every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours.
Effect of the Efferon LPS NEO hemoperfusion on the length of stay in the PICU | 1-14 days
  Time (number of days) from enrollment in the study to transfer from the PICU within 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Stepanenko, PhD, MD, Principal Investigator — Filatov Children's City Clinical Hospital of the Moscow Health Department; Igor Afukov, PhD, MD, Principal Investigator — Filatov Children's City Clinical Hospital of the Moscow Health Department
Locations (7):
- Russia (7):
  - Children's City Clinical Hospital named after St. Vladimir of the Moscow Department of Health, Moscow
  - Morozovskaya Children's City Clinical Hospital of the Moscow City Healthcare Department, Moscow
  - Clinical and Research Institute of Emergency Pediatric Surgery and Traumatology, Moscow
  - Filatov Children's City Clinical Hospital of the Moscow Health Department, Moscow
  - Children's City Clinical Hospital No. 9 named after G.N. Speransky of the Moscow City Health Department, Moscow
  - Children's City Clinical Hospital No. 5 named after N.F.Filatov, Saint Petersburg
  - Children's municipal multi-specialty clinical center of high medical technology, Saint Petersburg